CLINICAL TRIAL: NCT00569231
Title: A Phase 1 Study to Evaluate the Immunologic Mechanisms Underlying Wart Resolution After Intralesional Immunotherapy With Candida Antigen
Brief Title: Study With Candida Antigen for Treatment of Warts
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Allermed Laboratories, Inc. (Industry)
Responsible Party: Mayumi Nakagawa, University of Arkansas for Medical Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 46487
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Results first posted 2011-01-25 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2010-12

CONDITIONS: Warts; HPV
Keywords: Warts; Candida; HPV; Injections, Intralesional; Immune System
MeSH Terms: conditions — Warts; Torulopsis | interventions — PRA1 protein, Candida albicans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Candida Antigen (Experimental)
  Interventions: Drug: Candida Antigen

INTERVENTIONS:
Drug: Candida Antigen — Intralesional injection of 0.3ml candida antigen into largest wart at baseline visit and then every 3 weeks +/- 3 days for a maximum of 10 treatments.
  Other Names: Candin

SUMMARY:
The purpose of this study is to look at how people respond to the treatment of warts through use of the Candida antigen to get an immune response to rid the body of human papillomavirus (HPV). The immune system is the part of the body that fights infections like HPV which causes warts. This research study will examine the response of your wart when injected with a portion of a common yeast (candida) which is the study drug. Your immune system response will also be looked at by doing a test called an ELISPOT assay. This test is done on blood samples. The results of this test may help us to determine how the Candida antigen affects your wart.

DETAILED DESCRIPTION:
The use of recall antigens for treating warts is not yet Food and Drug Administration (FDA) approved. The primary goal of this work was to assess the safety of Candin as an investigational new drug (IND) for the treatment of warts. In addition, clinical resolution of treated and untreated warts was evaluated and immunologic responses were examined using an ex vivo interferon-γ enzyme-linked immunospot (IFN-γ ELISPOT) assay in order to elucidate the immunologic mechanisms behind the successful regression of warts in patients undergoing Candin injection immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be ages 18-50.
* Female subjects of child-bearing potential must have a negative urine pregnancy test before each treatment.
* Female subjects of child-bearing potential agree to use a reliable form of birth- control as the risks associated with candida antigens during pregnancy are not known.
* Subjects must have two or more cutaneous, non-genital, non-facial warts.
* Subjects must be able to provide written, informed consent.
* Subjects must be willing to comply with the requirements of the protocol.
* Subjects vital signs must be within the following parameters at time of enrollment:

  * Blood Pressure - <150/95 mmHg
  * Temperature - <100.4° F
  * Pulse Rate - 50 to 100 beats/minute
  * Respiratory Rate - <24 breaths/minute

Exclusion Criteria:

* Subjects who have a history of disease or treatment that has caused the subject to be immunosuppressed to include, but not limited to, cancer, HIV, or organ transplantation. Immunosuppression will be determined only by medical history.
* Subjects who are pregnant, lactating, or attempting to become pregnant, as the risks associated with candida antigens during pregnancy are not known.
* Subjects who have only genital or facial warts.
* Subjects who are unable to return for follow-up visits or comply with the protocol.
* Subjects who have a known allergy to Thimerosol or the candida antigen.
* Subjects who have a history of asthma as determined by a medical history or treatment for an asthmatic episode.
* Subjects who have any type of diabetes.
* Subjects who are currently using non-selective Beta Blockers.
* Subjects who are currently using H2 antagonists (e.g., cimetidine). There will be a 24 hour washout period for any use of H2 antagonists prior to beginning treatment in the study.
* Subjects who have a history of keloid formation.
* Subjects who have a history of alcohol or illicit drug abuse, as determined only by medical history.
* Subjects who have had previous treatment with candida antigens for their warts.
* Subjects who are currently using any other treatments for their warts. This includes prescription or over-the-counter medications. Subjects must have a wash¬out period of 30 days for any previous treatments prior to beginning the study.
* Subjects with a blood pressure >150/95, temperature >100.4° F, pulse rate <50 or >100 beats per minute, and respiratory rate >24 at time of enrollment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mayumi Nakagawa, MD, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Background] Majewski S, Jablonska S. Human papillomavirus-associated tumors of the skin and mucosa. J Am Acad Dermatol. 1997 May;36(5 Pt 1):659-85; quiz 686-8. doi: 10.1016/s0190-9622(97)80315-5. PMID 9146528
- [Background] Baker GE, Tyring SK. Therapeutic approaches to papillomavirus infections. Dermatol Clin. 1997 Apr;15(2):331-40. doi: 10.1016/s0733-8635(05)70441-1. PMID 9098642
- [Background] Miller DM, Brodell RT. Human papillomavirus infection: treatment options for warts. Am Fam Physician. 1996 Jan;53(1):135-43, 148-50. PMID 8546041
- [Background] Quan MB, Moy RL. The role of human papillomavirus in carcinoma. J Am Acad Dermatol. 1991 Oct;25(4):698-705. doi: 10.1016/0190-9622(91)70256-2. PMID 1665155
- [Background] Pfister H. Human papillomaviruses and skin cancer. Semin Cancer Biol. 1992 Oct;3(5):263-71. PMID 1335790
- [Background] MASSING AM, EPSTEIN WL. Natural history of warts. A two-year study. Arch Dermatol. 1963 Mar;87:306-10. doi: 10.1001/archderm.1963.01590150022004. No abstract available. PMID 13933441
- [Background] Johnson SM, Brodell RT. Treating warts: a review of therapeutic options. Consultant 1999;39(1):253-266.
- [Background] Brunk D. Injection of Candida antigen works on warts. Skin and Allergy News. 1999; 30(12):5.
- [Background] Johnson SM, Roberson PK, Horn TD. Intralesional injection of mumps or Candida skin test antigens: a novel immunotherapy for warts. Arch Dermatol. 2001 Apr;137(4):451-5. PMID 11295925
- [Background] Horn TD, Johnson SM, Helm RM, Roberson PK. Intralesional immunotherapy of warts with mumps, Candida, and Trichophyton skin test antigens: a single-blinded, randomized, and controlled trial. Arch Dermatol. 2005 May;141(5):589-94. doi: 10.1001/archderm.141.5.589. PMID 15897380
- [Derived] Coleman HN, Greenfield WW, Stratton SL, Vaughn R, Kieber A, Moerman-Herzog AM, Spencer HJ, Hitt WC, Quick CM, Hutchins LF, Mackintosh SG, Edmondson RD, Erickson SW, Nakagawa M. Human papillomavirus type 16 viral load is decreased following a therapeutic vaccination. Cancer Immunol Immunother. 2016 May;65(5):563-73. doi: 10.1007/s00262-016-1821-x. Epub 2016 Mar 15. PMID 26980480

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients for this study were recruited during the period between February 2007 and May 2009 from the outpatient Dermatology Clinic.
Groups:
- Candida Antigen: All patients enrolled into the study were treated with intralesional injection of 0.3ml candida antigen into largest wart at baseline visit and then every 3 weeks +/- 3 days for a maximum of 10 treatments.
Period: Overall Study
Arm/Group | Candida Antigen
Started | 18
Completed | 11
Not Completed | 7
Not completed — Study unrelated surgery | 1
Not completed — Airfare expense | 2
Not completed — Withdrawal by Subject | 1
Not completed — Car accident injury | 1
Not completed — Non-compliance | 2

BASELINE CHARACTERISTICS:
Arm/Group | Candida Antigen
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 29.8 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Resolution of Injected Wart
Description: When the participant completed the protocol, clinical resolution of the injected wart was determined by the overall percentage of resolution from the initial visit. Participants were classified as 'complete responders' if they had complete resolution of the injected wart, 'partial responders' if the injected wart regressed between 25% and 99%, and 'non-responders' if they had not achieved at least 25% regression of the injected wart.
Time Frame: Initial visit to completion of protocol, which is up to 30 weeks
Population: The participants were analyzed if they completed the protocol by achieving complete resolution of the treated wart, receiving the maximum of 10 treatments, or by having less than 25% resolution of the treated wart after 5 treatments.
Measure: Number; unit: Participants
Arm/Group | Candida Antigen
Number analyzed (Participants) | 11
Participants
  Complete responder | 9
  Partial responder | 1
  Non-responder | 1

2. Secondary Outcome: Number of Participants With Clinical Resolution of 1st Anatomically Distant, Non-injected Wart
Description: When the participant completed the protocol, clinical resolution of 1st anatomically distant, non-injected wart was determined by the overall percentage of resolution from the initial visit.
Time Frame: Initial visit to completion of protocol, which is up to 30 weeks
Population: Participants with 1st anatomically distant, non-injected wart were analyzed.
Measure: Number; unit: Participants
Arm/Group | Candida Antigen
Number analyzed (Participants) | 8
Participants
  Complete resolution of 1st non-injected wart | 6
  Partial resolution of 1st non-injected wart | 2

3. Secondary Outcome: Number of Participants With Clinical Resolution of 2nd Anatomically Distant, Non-injected Wart
Description: When the participant completed the protocol, clinical resolution of 2nd anatomically distant, non-injected wart was determined by the overall percentage of resolution from the initial visit.
Time Frame: Initial visit to completion of protocol, which is up to 30 weeks
Population: The participants with 2nd anatomically distant, non-injected wart were analyzed.
Measure: Number; unit: Participants
Arm/Group | Candida Antigen
Number analyzed (Participants) | 6
Participants | 6

4. Other Pre Specified Outcome: Number of Participants With Immune Response to Human Papillomavirus Type 57 (HPV-57) L1-peptide
Description: Immunologic responses from peripheral blood mononuclear cells collected prior to vaccination and post-vaccination were measured by ex vivo interferon-γ enzyme-linked immunospot (IFN-γ ELISPOT) assay to human papillomavirus type 57 L1-peptide.
Time Frame: Initial visit to completion of protocol, which is up to 30 weeks
Population: The interferon-γ enzyme-linked immunospot assay was performed on available samples from participants who completed the study.
Measure: Number; unit: Participants
Arm/Group | Candida Antigen
Number analyzed (Participants) | 10
Participants | 6

ADVERSE EVENTS:
Time Frame: 3 years, 4 months
Arm/Group | Candida Antigen
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 15/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Candida Antigen (N=18)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Chills (General disorders) | 1 (1) — Vaccine-unrelated adverse event
Flu like symptoms (General disorders) | 2 (3)
Headache (Nervous system disorders) | 2 (3)
Hematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) — Vaccine-unrelated adverse event.
Injection site reaction (General disorders) | 15 (74)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (3) — Vaccine-unrelated adverse event
Lymph node pain (Blood and lymphatic system disorders) | 1 (2)
Malaise (General disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes